CLINICAL TRIAL: NCT02763059
Title: Comparison Between Dexamethasone and Ibuprofen on Postoperative Pain Prevention and Control Following Surgical Implant Placement: a Double-Blind, Parallel-Group, Placebo-Controlled Randomized Clinical Trial
Brief Title: Comparison Between Dexamethasone and Ibuprofen on Pain Prevention and Control Following Surgical Implant Placement
Acronym: CBDIPPCFSIP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Maha A. Bahammam, Associate Professor and Consultant of Periodontology, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1434/254/287
Record Dates: First submitted 2016-05-01; First posted 2016-05-05 (Estimated); Results first posted 2025-10-29 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Pain Measurement
MeSH Terms: interventions — Ibuprofen; Dexamethasone; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1- Received Ibuprofen (N=44) (Active Comparator): This group receives 1 hour before surgery 600 mg ibuprofen (and another 600 mg dose 6 hours after the first dose).
  Acetaminophen 1000 mg: A Rescue medication (1000 mg acetaminophen) was given to each patient who was instructed to take it if necessary.
  Interventions: Drug: Ibuprofen 600 mg; Drug: Acetaminophen 1000 mg
- Group 2- Received Dexamethasone (N=44) (Active Comparator): This group receives 1 hour before surgery 4 mg dexamethasone (and another 4 mg 6 hours after the first dose) Acetaminophen 1000 mg: A Rescue medication (1000 mg acetaminophen) was given to each patient who was instructed to take it if necessary.
  Interventions: Drug: Dexamethasone 4 mg; Drug: Acetaminophen 1000 mg
- Group 3 - Received Placebo (N=44) (Placebo Comparator): This group receives 1 hour before surgery placebo. Acetaminophen 1000 mg: A Rescue medication (1000 mg acetaminophen) was given to each patient who was instructed to take it if necessary.
  Interventions: Drug: Placebo; Drug: Acetaminophen 1000 mg

INTERVENTIONS:
Drug: Ibuprofen 600 mg — This group receives 1 hour before surgery 600 mg ibuprofen (and another 600 mg dose 6 hours after the first dose);
  Other Names: 600 mg ibuprofen (and another 600 mg dose 6 hours after the first dose).
  Arms: Group 1- Received Ibuprofen (N=44)
Drug: Dexamethasone 4 mg — This group receives 1 hour before surgery 4 mg dexamethasone (and another 4 mg 6 hours after the first dose)
  Other Names: 4 mg dexamethasone (and another 4 mg 6 hours after the first dose)
  Arms: Group 2- Received Dexamethasone (N=44)
Drug: Placebo — This group receives 1 hour before surgery placebo.
  Other Names: Acetaminophen 1000 mg
  Arms: Group 3 - Received Placebo (N=44)
Drug: Acetaminophen 1000 mg — A Rescue medication (1000 mg acetaminophen) was given to each patient who was instructed to take it if necessary.
  Other Names: A Rescue medication (1000 mg acetaminophen) was given to each patient who was instructed to take it if necessary.

SUMMARY:
Background and aim: Postoperative pain is an adverse effect of oral surgeries and may therefore be prevented or minimized. This study compares the efficacy of preemptive ibuprofen and dexamethasone protocols in pain prevention and control after surgical implant placement.

Methods: For this prospective, double-masked, parallel-group, placebo-controlled, randomized clinical trial, 117 dental implants were placed. The groups received three different protocols 1 hour before surgery:

1. 600 mg ibuprofen (and another 600 mg dose 6 hours after the first dose);
2. 4 mg dexamethasone (and another 4 mg 6 hours after the first dose) or
3. placebo.

Rescue medication (1000 mg acetaminophen) was given to each patient who was instructed to take it if necessary. Pain intensity was evaluated by a 101-point numeric rate scale and visual analogue scale, additionally discomfort was evaluated using a four-point verbal rate scale, hourly for the first 8 hours after surgery and three times a day on the following 3 days.

DETAILED DESCRIPTION:
This prospective clinical trial investigated the efficacy of preemptive medication in mitigating postoperative pain following dental implant surgeries. With a sample size of 117 participants, the study employed a double-masked, parallel-group, placebo-controlled design. Patients were randomly assigned to receive one of three treatment protocols-an ibuprofen regimen, a dexamethasone regimen, or a placebo-administered one hour before surgery. Pain intensity and discomfort were assessed using numeric, visual, and verbal scales hourly for the first 8 hours post-surgery, followed by thrice-daily evaluations for the next 3 days. Additionally, rescue medication (acetaminophen) was provided to manage pain as needed. The study aimed to determine whether ibuprofen or dexamethasone could effectively alleviate postoperative pain compared to a placebo to highlight optimal pain management strategies for dental implant procedures.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent for the described procedure
* Surgical placement of a single endosteal implant
* Age of at least 18 years

Exclusion Criteria:

* The need for bone grafting or sinus lift for implant placement
* Pregnant and lactating women
* Metabolic disorders
* Immunocompromised status
* Hemophilia or bleeding disorders
* Drug or alcohol abuse
* Treatment with steroids in the previous 6 months
* History of radiation therapy in the head and neck
* Psychiatric disorders
* Inability to understand the procedure described in the questionnaire

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2013-09; Primary Completion 2015-05 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maha Bahammam, Sc, CAGS, EdM, DABP, Study Director — King Abdulaziz University

REFERENCES:
- [Derived] Bahammam MA, Kayal RA, Alasmari DS, Attia MS, Bahammam LA, Hassan MH, Alzoman HA, Almas K, Steffens JP. Comparison Between Dexamethasone and Ibuprofen for Postoperative Pain Prevention and Control After Surgical Implant Placement: A Double-Masked, Parallel-Group, Placebo-Controlled Randomized Clinical Trial. J Periodontol. 2017 Jan;88(1):69-77. doi: 10.1902/jop.2016.160353. Epub 2016 Aug 26. PMID 27562219

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1- Received Ibuprofen (N=44) | Group 2- Received Dexamethasone (N=44) | Group 3 - Received Placebo (N=44)
Started | 44 | 44 | 44
Completed | 39 | 43 | 35
Not Completed | 5 | 1 | 9
Not completed — Lost to Follow-up | 4 | 1 | 6
Not completed — Withdrawal by Subject | 1 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Group 1- Received Ibuprofen (N=39): Ibuprofen 600 mg: This group receives 1 hour before surgery 600 mg ibuprofen (and another 600 mg dose 6 hours after the first dose);
  Acetaminophen 1000 mg: A Rescue medication (1000 mg acetaminophen) was given to each patient who was instructed to take it if necessary.
- Group 2- Received Dexamethasone (N=43): Dexamethasone 4 mg: This group receives 1 hour before surgery 4 mg dexamethasone (and another 4 mg 6 hours after the first dose)
  Acetaminophen 1000 mg: A Rescue medication (1000 mg acetaminophen) was given to each patient who was instructed to take it if necessary.
- Group 3 - Received Placebo (N=35): Placebo: This group receives 1 hour before surgery placebo.
  Acetaminophen 1000 mg: A Rescue medication (1000 mg acetaminophen) was given to each patient who was instructed to take it if necessary.
- Total: Total of all reporting groups
Arm/Group | Group 1- Received Ibuprofen (N=39) | Group 2- Received Dexamethasone (N=43) | Group 3 - Received Placebo (N=35) | Total
Number analyzed (Participants) | 39 | 43 | 35 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 43 | 35 | 117
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] — Inclusion criteria
  1. written informed consent for the described procedure;
  2. surgical placement of a single endosteal implant; and
  3. age >18 years.
  years | 33.0 [32.0 to 37.0] | 35.0 [33.0 to 44.0] | 41.0 [34.0 to 50.0] | 35 [32.0 to 50.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 23 | 20 | 54
  Male | 28 | 20 | 15 | 63
Region of Enrollment [Number; unit: participants]
  Saudi Arabia | 39 | 43 | 35 | 117

OUTCOME MEASURES:

1. Primary Outcome: The Visual Analog Scale (VAS) Was Used to Measures Levels of Pain.
Description: The Visual Analog Scale (VAS) is a 10-cm line with two extremes at either end: "no pain" (0) and "pain that could not be more severe" (10). Patients were asked to mark a point on the line that best represented their perceived level of pain. The marked position on the line was then measured in centimeters to provide a score between 0 and 10.
  * Minimum Score: 0 (No pain)
  * Maximum Score: 10 (Pain that could not be more severe)
  * Interpretation: Lower scores indicate better outcomes, representing lower levels of perceived pain. Higher scores indicate worse outcomes, representing greater levels of pain.
  * Unit of Measure: Scores on a scale (0-10)
Time Frame: 8 hours-time
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group 1- Received Ibuprofen (N=39) | Group 2- Received Dexamethasone (N=43) | Group 3 - Received Placebo (N=35)
Number analyzed (Participants) | 39 | 43 | 35
score on a scale | 2 [1.08 to 4.40] | 2 [1.57 to 3.00] | 5.0 [3.96 to 7.01]

2. Secondary Outcome: the 101-point Numerical Rate Scale (NRS-101) Was Used to Measures Levels of Pain.
Description: The Numerical Rating Scale (NRS-101) is a scale ranging from 0 to 100, where 0 represents "no pain" and 10(0) represents either "the worst possible pain" or "the most intense pain imaginable".
  * Minimum Score: 0 (No pain)
  * Maximum Score: 100 (Worst possible pain)
  * Interpretation: Lower scores indicate better outcomes, representing lower levels of perceived pain. Higher scores indicate worse outcomes, representing higher levels of perceived pain.
  * Unit of Measure: Scores on a scale (0-100)
Time Frame: 8 hours-time
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Group 1- Received Ibuprofen (N=39) | Group 2- Received Dexamethasone (N=43) | Group 3 - Received Placebo (N=35)
Number analyzed (Participants) | 39 | 43 | 35
score on a scale | 5 [4.74 to 9.19] | 6 [5.66 to 8.37] | 39 [33.65 to 45.06]

3. Secondary Outcome: The 4-point Verbal Rating Scale (VRS-4) Was Used to Measures Levels of Discomfort.
Description: The 4-point Verbal Rating Scale (VRS-4) is a verbal scale used to assess the severity of a given condition, such as pain. Patients rate their experience by selecting one of four verbal descriptors that best represents their perceived intensity, ranging from "no pain" to "severe pain."
  * Minimum Score: 0 (No pain)
  * Maximum Score: 3 (Severe pain)
  * Interpretation: Lower scores indicate better outcomes, representing lower levels of perceived severity. Higher scores indicate worse outcomes, representing greater levels of severity.
  * Unit of Measure: Scores on a scale (0-3)
Time Frame: 8 hours-time
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Group 1- Received Ibuprofen (N=39) | Group 2- Received Dexamethasone (N=43) | Group 3 - Received Placebo (N=35)
Number analyzed (Participants) | 39 | 43 | 35
score on a scale | 1 [1 to 1] | 1 [1 to 1] | 2 [1 to 3]
Statistical Analysis 1: Comparison: Group 1- Received Ibuprofen (N=39) vs Group 2- Received Dexamethasone (N=43) vs Group 3 - Received Placebo (N=35); The Kruskal-Wallis test is an omnibus test comparing all three independent groups; Test type: Other — Kruskal-Wallis; p = 0.027, Kruskal-Wallis — Kruskal-Wallis test, a non-parametric omnibus test, was used followed by Dunn's multiple comparison test for pairwise group analysis. A priori threshold for statistical significance was set at p < 0.05 with no adjustments for multiple comparisons
Statistical Analysis 2: Comparison: Group 1- Received Ibuprofen (N=39) vs Group 2- Received Dexamethasone (N=43) vs Group 3 - Received Placebo (N=35); The Kruskal-Wallis test is an omnibus test comparing all three independent groups on the pain/discomfort outcome; Test type: Other — Kruskal-Wallis; p < 0.0001, Kruskal-Wallis — [p-value comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Arm/Group | Group 1- Received Ibuprofen (N=39) | Group 2- Received Dexamethasone (N=43) | Group 3 - Received Placebo (N=35)
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/43 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/43 | 0/35
Other Adverse Events (participants affected / at risk) | 0/39 | 0/43 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes